CLINICAL TRIAL: NCT01114659
Title: The Study of Metabolic and Cardiac Vascular Risk in Patients With Polycystic Ovary Syndrome
Brief Title: The Study of Polycystic Ovary Syndrome(PCOS) With Gene and Questionnaire
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Ming-I Hsu, MD, Attending Doctor, Taipei Medical University WanFang Hospital
Other Study IDs: WFH-PCOS-98076
Record Dates: First submitted 2010-04-29; First posted 2010-05-03 (Estimated); Last update posted 2014-01-01 (Estimated); Status verified 2013-12

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Women with PCOS
- Normal Control

SUMMARY:
Polycystic ovary syndrome (PCOS) is an extremely common disorder in women of reproductive age. Diagnosis of PCOS is principally based on clinical and physical findings. Diagnostic criteria and PCOS definitions used by clinicians and researchers are almost as heterogeneous as the syndrome. This first part of study is determine whether genetic polymorphisms influence hormonal and metabolic characteristics in Taiwanese patients with PCOS and controls. Furthermore, women with PCOS were reported with high risk of cardiovascular disease, the investigators planned to calculate the difference of carotid intima-media thickness (IMT) and B-type natriuretic peptide (BNP) between women with PCOS and normal control to determine the premature atherosclerosis of women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* women at reproductive age
* women with PCOS and women without PCOS.

Exclusion Criteria:

* young women who had their menarche less than 3 years
* women older than 45 years old, Amenorrhea of menopause, hyperglycemia, hyperthyroidism, hypothyroidism, heart failure, lung failure, renal failure, anemia, dystrophy, gonitis.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Polycystic Ovary Syndrome(PCOS)
Sampling Method: Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2009-11; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The correlation of PCOS betwwen metabolic and cardiovascular disease. | Participant were followed for 1 month in study period.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-I Hsu, MD, Principal Investigator — Wan Fang Hospital
Locations (1):
- Taipei Medical University WanFang Hospital, Taipei, Taipei, Taiwan